CLINICAL TRIAL: NCT00002525
Title: Phase III Intergroup Prospectively Randomized Trial of Perioperative 5-FU After Curative Resection, Followed by 5-FU/Leucovorin for Patients With Colon Cancer
Brief Title: Perioperative Chemotherapy in Treating Patients With Colon Cancer That Can Be Surgically Removed
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped before reaching its accrual goal due to slow accrual
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network); Cancer and Leukemia Group B (Network); American College of Surgeons (Other); NSABP Foundation Inc (Network)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E1292; E1292 (Other: ECOG-ACRIN Cancer Research Group); U10CA023318 (NIH); CDR0000078337 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 1999-11-01; First posted 2004-04-06 (Estimated); Results first posted 2016-07-20 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; stage III colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perioperative 5-FU (Experimental): Within 24 hours of the colon resection, patients receive perioperative fluorouracil intravenously (IV) over 24 hours for 7 days.
  After surgery (beginning 21-35 days post-surgery), 5-FU was given at a dose of 425 mg/m^2 IV push on days 1-5, and leucovorin calcium was given at a dose of 20mg/m^2 IV push on days 1-5
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium
- No perioperative 5-FU (Active Comparator): Patients receive no perioperative fluorouracil.
  After surgery (beginning 21-35 days post-surgery), 5-FU was given at a dose of 425 mg/m^2 IV push on days 1-5, and leucovorin calcium was given at a dose of 20mg/m^2 IV push on days 1-5
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium

INTERVENTIONS:
Drug: fluorouracil — Perioperative 5-FU: 600 mg/m^2/d x 7 days continuous IV, beginning within 24 hours of surgery
  After surgery, 5-FU was given 425 mg/m^2 IV push on days 1-5
  Other Names: 5-FU; Adrucil; Efudex
Drug: leucovorin calcium — given after surgery at dose of 20mg/m^2 IV push on days 1-5
  Other Names: Leucovorin; Wellcovorin; Citrovorum factor; Folinic acid; 5-formyl tetrahydrofolate; LV; LCV

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving drugs in different ways may kill more tumor cells. It is not yet known if surgery is more effective with or without chemotherapy for colon cancer.

PURPOSE: Randomized phase III trial to evaluate whether perioperative 5-Fluorouracil (5-FU) chemotherapy after curative resection could improve overall survival and disease-free survival in patients with Duke's B3 or C colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine if adjuvant therapy with one week of continuous 5-FU given within 24 hours of a curative colon resection followed by 6 months of 5-FU/leucovorin is effective in prolonging the disease-free survival and increasing overall survival in patients with Dukes' B3 or C colon cancer, when compared to patients who are treated with 5-FU/leucovorin only.

II. 1. To determine if a week of perioperative continuous 5-FU affects disease-free survival and overall survival in patients with Dukes' B2 colon cancer.

OUTLINE: This is an open-label, randomized phase III study. Patients undergo curative colon resection via laparotomy. Patients are randomized to 1 of 2 arms in a 1:1 ratio.

Arm I (Perioperative 5-FU): Within 24 hours of the colon resection, patients receive perioperative 5-fluorouracil (5-FU) intravenously (IV) over 24 hours for 7 days.

Arm II (No perioperative 5-FU): Patients receive no perioperative fluorouracil.

After surgery, patients with stage I, stage IIA, or stage IV colon cancer are immediately removed from study. Patients with stage IIB, IIC, or III colon cancer are re-registered within 35 days postoperatively. Beginning 21-35 days after surgery, patients with stage IIC or III disease receive leucovorin calcium IV bolus immediately followed by 5-FU IV bolus on days 1-5. Courses repeat every 28 days for a total of 6 courses in the absence of disease progression or unacceptable toxicity. Patients with stage IIB disease do not receive adjuvant 5-FU and leucovorin calcium.

Patients are followed every 3 months for 2 years, then every 6 months for 2 years, and then annually until 15 years.

PROJECTED ACCRUAL: A total of 800-2,000 patients (at least 400 per treatment arm) will be accrued for this study over 2-3 years.

ELIGIBILITY:
Eligibility Criteria for Randomization:

Inclusion Criteria:

* Adenocarcinoma of the colon documented by colonoscopy or barium enema
* Tumor either considered resectable or totally resected within 24 hours prior to study
* Randomization within 2 weeks prior to surgery or within 24 hours after surgery required
* Patients randomized after surgery must meet the following criteria:

  * Complete resection performed with no evidence of residual disease or distant metastases
  * Distal margin of tumor above the peritoneal reflection in area of rectum
  * No free perforation Intestinal obstruction allowed
  * Preliminary or complementary colostomy allowed
* Concurrent registration for E3293 strongly recommended
* Age 18 and over
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Adequate organ function based on the following tests within 2 weeks prior to randomization

  * White Blood Cell (WBC) at least 3,000/mm^3
  * Platelet count at least 100,000/mm^3
  * Bilirubin no greater than 2.0 mg/dL
  * Creatinine no greater than 2.0 mg/dL
* No second malignancy within 5 years except: superficial non-melanomatous skin cancer and carcinoma in situ of the cervix
* Fertile patients must use adequate contraception

Exclusion Criteria:

* Dual primary tumors
* Prior nonmalignant systemic disease that would preclude use of chemotherapy
* Pregnant or nursing
* Prior fluorouracil
* Other prior or concurrent chemotherapy for this malignancy
* Prior or concurrent radiotherapy for this malignancy

Eligibility Criteria for Re-registration for Patients Randomized Pre-operatively:

* Must have pathologic classification of Dukes' B2, B3, or C disease by the contributing institution.
* Must be re-registered < 35 days after surgery.
* ECOG performance status of 0-2.
* Complete resection must have been performed with no evidence of residual disease or distant metastasis.
* Distal margin of the tumor must not extend below the peritoneal reflection in the area of the rectum.
* Single primary colon carcinoma without free perforation demonstrated. Patients with intestinal obstruction are eligible. Preliminary or complementary colostomy dose not preclude entry of a patient.
* Have WBC > 3000/mm^3, platelets > 100,000/mm^3, adequate renal (serum creatinine <= 2.0mg/dL) and hepatic function (bilirubin <= 2.0mg/dL), within one week prior to beginning adjuvant chemotherapy (For Dukes' B3 and C patients only).

Eligibility Criteria for Re-registration for Patients Randomized Post-operatively:

* Must have pathologic classification of Dukes' B2, B3, or C disease by the contributing institution.
* Patient must be re-registered < 35 days after surgery.
* ECOG performance status of 0-2.
* Started perioperative 5-FU, if assigned, within 24 hours of surgery.
* Have WBC > 3000/mm^3, platelets > 100,000/mm^3, adequate renal (serum creatinine <= 2.0mg/dL) and hepatic function (bilirubin < =2.0mg/dL), within one week prior to beginning adjuvant chemotherapy (For Dukes' B3 and C patients only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 859 (Actual)
Dates: Start 1993-10-01 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary M. Kemeny, MD, FACS, Study Chair — SUNY at Stony Brook
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Result] Kemeny M, Ibrahim J, Benson AB, et al.: Post-operative complications of continuous infusion 5 FU following curative resection of colon cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 16: A923, 260a, 1997.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on August 20, 1993 and was terminated on May 19, 2000 before reaching its accrual goal due slow accrual. The first accrual was on October 1, 1993. The final accrual for the study was 859 patients.
Groups:
- Perioperative 5-FU: Within 24 hours of the colon resection, patients receive perioperative fluorouracil intravenously (IV) over 24 hours for 7 days.
  After surgery (beginning 21-35 days post-surgery), 5-FU was given at a dose of 425 mg/m^2 IV push on days 1-5, and leucovorin calcium was given at a dose of 20mg/m^2 IV push on days 1-5
  fluorouracil: Perioperative 5-FU: 600 mg/m^2/d x 7 days continuous IV, beginning within 24 hours of surgery
  After surgery, 5-FU was given 425 mg/m^2 IV push on days 1-5
  leucovorin calcium: given after surgery at dose of 20mg/m^2 IV push on days 1-5
- No Perioperative 5-FU: Patients receive no perioperative fluorouracil.
  After surgery (beginning 21-35 days post-surgery), 5-FU was given at a dose of 425 mg/m^2 IV push on days 1-5, and leucovorin calcium was given at a dose of 20mg/m^2 IV push on days 1-5 fluorouracil: Perioperative 5-FU: 600 mg/m^2/d x 7 days continuous IV, beginning within 24 hours of surgery After surgery, 5-FU was given 425 mg/m^2 IV push on days 1-5 leucovorin calcium: given after surgery at dose of 20mg/m^2 IV push on days 1-5
Period: Overall Study
Arm/Group | Perioperative 5-FU | No Perioperative 5-FU
Started | 427 (859 patients were enrolled to the study, but 4 patients were not randomized to any treatment arm) | 428
Treated | 419 | 0 (Patients on "No perioperative 5-FU arm" received no perioperative chemotherapy)
Dukes' B3 or C Stage | 156 (Primary population: pts with Duke's B3, C disease. 158 such pts on "No perioperative 5-FU arm") | 158
Dukes' B2 Stage | 150 | 139
Completed | 241 | 428 (Patients on "No perioperative 5-FU arm" received no perioperative chemotherapy)
Not Completed | 186 | 0
Not completed — Adverse Event | 36 | 0
Not completed — Death | 5 | 0
Not completed — Withdrawal by Subject | 11 | 0
Not completed — Start non-protocol therapy | 1 | 0
Not completed — Other complicating disease | 1 | 0
Not completed — Duke's A, B1, D disease | 92 | 0
Not completed — Error | 6 | 0
Not completed — Other | 26 | 0
Not completed — Never start protocol therapy | 8 | 0

BASELINE CHARACTERISTICS:
Population: The primary analysis population for the study was all randomized patients with Duke's B3 and C disease.
Groups:
- Total: Total of all reporting groups
Arm/Group | Perioperative 5-FU | No Perioperative 5-FU | Total
Number analyzed (Participants) | 156 | 158 | 314
Age, Continuous [Median (Full Range); unit: Years] | 63 [30 to 89] | 66 [25 to 86] | 65 [25 to 89]
Sex/Gender, Customized [Number; unit: participants] — 1 patient on "No perioperative 5-FU arm" had missing information about sex
  participants
    Female | 57 | 61 | 118
    Male | 99 | 96 | 195

OUTCOME MEASURES:

1. Primary Outcome: 5-year Overall Survival Rate in Patients With Dukes' B3/C Disease
Description: Overall survival (OS) is defined as time from randomization to death from any cause or last date known alive. Kaplan-Meier method was used to estimate 5-year OS rate
Time Frame: every 3 months for 2 years, then every 6 months for 2 years, and then annually until year 15 after randomization
Population: All randomized patients with Dukes' B3 and C disease
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Perioperative 5-FU | No Perioperative 5-FU
Number analyzed (Participants) | 156 | 158
proportion of participants | 0.666 [0.585 to 0.735] | 0.612 [0.530 to 0.683]
Statistical Analysis 1: Comparison: Perioperative 5-FU vs No Perioperative 5-FU; Test type: Superiority or Other; p = 0.178, Log Rank — one-sided log-rank test p value

2. Secondary Outcome: 5-year Disease-free Survival Rate in Patients With Dukes' B3/C Disease
Description: Disease-free survival (DFS) was defined as time from randomization to recurrence, second invasive primary cancer, or deaths, whichever occurred first. Patients who were still alive and had no DFS events were censored at the last disease assessment date known to be free of DFS events. Patients without any follow up data were censored at random assignment. Kaplan-Meier method was used to estimate the 5-year DFS rate.
Time Frame: every 3 months for 2 years, then every 6 months for 2 years, and then annually until year 15 after randomization
Population: All randomized patients with Dukes' B3 and C disease who had complete disease assessment data
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Perioperative 5-FU | No Perioperative 5-FU
Number analyzed (Participants) | 128 | 131
proportion of participants | 0.582 [0.486 to 0.668] | 0.543 [0.442 to 0.634]
Statistical Analysis 1: Comparison: Perioperative 5-FU vs No Perioperative 5-FU; Test type: Superiority or Other; p = 0.847, Log Rank — two-sided log rank test

3. Secondary Outcome: 5-year Overall Survival Rate in Patients With Dukes' B2 Disease
Description: as for outcome 1
Time Frame: every 3 months for 2 years, then every 6 months for 2 years, and then annually until year 15 after randomization
Population: All randomized patients with Dukes' B2 disease
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Perioperative 5-FU | No Perioperative 5-FU
Number analyzed (Participants) | 150 | 139
proportion of participants | 0.851 [0.783 to 0.899] | 0.780 [0.701 to 0.841]

4. Secondary Outcome: 5-year Disease-free Survival Rate in Patients With Dukes' B2 Disease
Description: as for outcome 2
Time Frame: every 3 months for 2 years, then every 6 months for 2 years, and then annually until year 15 after randomization
Population: All randomized patients with Dukes' B2 disease who had complete disease assessment data
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Perioperative 5-FU | No Perioperative 5-FU
Number analyzed (Participants) | 133 | 123
proportion of participants | 0.749 [0.660 to 0.818] | 0.724 [0.626 to 0.801]

ADVERSE EVENTS:
Time Frame: Patients on Arm I received perioperative 5-FU, patients on Arm II received no perioperative chemotherapy. AEs, however, were reported for all patients and assessed at the end of treatment and 30 days after the last dose of the therapy.
Description: After completion of perioperative 5-FU, patients with Dukes' B3/C disease continued to receive the then standard adjuvant chemotherapy for colon cancer. AEs for the adjuvant chemotherapy (5-FU+ Levamisolem and 5-FU+Leucovovin) in patients with Dukes' B3/C disease were collected separately and reported here as well.
Groups:
- Arm I (Perioperative 5-FU): Within 24 hours of the colon resection, patients receive perioperative fluorouracil intravenously (IV) over 24 hours for 7 days.
  After surgery (beginning 21-35 days post-surgery), 5-FU was given at a dose of 425 mg/m^2 IV push on days 1-5, and leucovorin calcium was given at a dose of 20mg/m^2 IV push on days 1-5
  fluorouracil: Perioperative 5-FU: 600 mg/m^2/d x 7 days continuous IV, beginning within 24 hours of surgery
  After surgery, 5-FU was given 425 mg/m^2 IV push on days 1-5
  leucovorin calcium: given after surgery at dose of 20mg/m^2 IV push on days 1-5
- Arm II (No Perioperative 5-FU): Patients receive no perioperative fluorouracil.
  After surgery (beginning 21-35 days post-surgery), 5-FU was given at a dose of 425 mg/m^2 IV push on days 1-5, and leucovorin calcium was given at a dose of 20mg/m^2 IV push on days 1-5
  fluorouracil: Perioperative 5-FU: 600 mg/m^2/d x 7 days continuous IV, beginning within 24 hours of surgery
  After surgery, 5-FU was given 425 mg/m^2 IV push on days 1-5
  leucovorin calcium: given after surgery at dose of 20mg/m^2 IV push on days 1-5
- Adjuvant Chemotherapy-- 5-FU+Levamisolem: Beginning 21-35 days after surgery, patients with stage IIC or III disease enrolled between September 1997 and May 2000 receive the following adjuvant chemotherapy:
  Leucovorin: 20 mg/m² IV push days 1-5 5-FU: 425 mg/m² IV push days 1-5, give immediately after Leucovorin
  A cycle of therapy consisted of 5 consecutive days of chemotherapy. Cycles were repeated at the end of 4 weeks (day 29), 8 weeks (day 57) and then every 4 weeks for a total of 6 cycles.
  All patients with Dukes' B3/C disease for who adverse vents were collected were included in the analysis.
- Adjuvant Chemotherapy-- 5-FU+Leucovovin: After surgery, patients with stage IIC or III disease enrolled between August 1993 and August 1997 receive the following adjuvant chemotherapy:
  Levamisole: 50 mg PO TID Days 1-3 and Days 15-17; 50 mg PO TID x 3 days beginning Day 29, repeat every 14 days for 11 months.
  5-FU: 450 mg/m²/day IV bolus for Days 1-5. 450 mg/m² IV bolus once weekly beginning Day 29, repeat weekly for a maximum of 11 months.
  All patients with Dukes' B3/C disease for who adverse vents were collected were included in the analysis.
Arm/Group | Arm I (Perioperative 5-FU) | Arm II (No Perioperative 5-FU) | Adjuvant Chemotherapy-- 5-FU+Levamisolem | Adjuvant Chemotherapy-- 5-FU+Leucovovin
Serious Adverse Events (participants affected / at risk) | 75/418 | 4/422 | 76/171 | 32/61
Other Adverse Events (participants affected / at risk) | 236/418 | 9/422 | 167/171 | 58/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Perioperative 5-FU) (N=418) | Arm II (No Perioperative 5-FU) (N=422) | Adjuvant Chemotherapy-- 5-FU+Levamisolem (N=171) | Adjuvant Chemotherapy-- 5-FU+Leucovovin (N=61)
Leukopenia (Investigations) | 3 | 1 | 23 | 8
Granulocytopenia (Investigations) | 1 | 0 | 4 | 1
Anemia (Blood and lymphatic system disorders) | 22 | 0 | 1 | 1
Infection (Infections and infestations) | 9 | 0 | 1 | 3
Nausea/Vomiting (Gastrointestinal disorders) | 7 | 0 | 8 | 4
Vomiting (Gastrointestinal disorders) | 6 | 0 | 5 | 2
Diarrhea (Gastrointestinal disorders) | 14 | 0 | 20 | 15
Stomatitis (Gastrointestinal disorders) | 11 | 0 | 6 | 9
Liver (Hepatobiliary disorders) | 2 | 0 | 5 | 1
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 1
Cardiac (Cardiac disorders) | 9 | 0 | 2 | 2
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0
Skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 3
Neuro-sensory (Nervous system disorders) | 0 | 1 | 3 | 0
Neuro-motor (Nervous system disorders) | 6 | 0 | 1 | 4
Neuro-psych (Nervous system disorders) | 1 | 0 | 3 | 1
Others (General disorders) | 0 | 2 | 7 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Phlebitis (Blood and lymphatic system disorders) | 0 | 0 | 5 | 2
Neuro-clinical (Nervous system disorders) | 0 | 0 | 6 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Perioperative 5-FU) (N=418) | Arm II (No Perioperative 5-FU) (N=422) | Adjuvant Chemotherapy-- 5-FU+Levamisolem (N=171) | Adjuvant Chemotherapy-- 5-FU+Leucovovin (N=61)
Leukopenia (Investigations) | 25 | 2 | 78 | 32
Thrombocytopenia (Investigations) | 24 | 0 | 66 | 14
Anemia (Blood and lymphatic system disorders) | 209 | 7 | 105 | 43
Fever (No Infection) (General disorders) | 45 | 1 | 15 | 7
Nausea/vomiting (Gastrointestinal disorders) | 116 | 4 | 94 | 27
Vomiting (Gastrointestinal disorders) | 60 | 3 | 45 | 11
Diarrhea (Gastrointestinal disorders) | 67 | 3 | 74 | 27
Stomatitis (Gastrointestinal disorders) | 71 | 1 | 59 | 20
Skin (Skin and subcutaneous tissue disorders) | 39 | 2 | 73 | 24
Neuro-clinical (Nervous system disorders) | 21 | 1 | 84 | 18
Infection (Infections and infestations) | 0 | 0 | 33 | 9
Neuro-motor (Nervous system disorders) | 6 | 0 | 33 | 3
Neuro-psych (Nervous system disorders) | 9 | 1 | 17 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less